CLINICAL TRIAL: NCT01076777
Title: Effects of Physical Exercise on Anxiety and Co-morbid Emotional Disturbances: A Clinical Trail in a Day Care Unit
Brief Title: Physical Exercise Versus Cognitive-behavioral Therapy (CBT) for Panic Disorders: A Randomised Controlled Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Norwegian Department of Health and Social Affairs (Other Government)
Responsible Party: Professor Inger Hilde Nordhus, Faculty of Psychology at University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3.2007.499 (REK)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Panic Disorder
Keywords: Panic disorder; Physical exercise; Cognitive-behavioral therapy; Manualized
MeSH Terms: conditions — Panic Disorder; Motor Activity | interventions — Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical exercise (Experimental): Manualised Exercise performed in groups (5-8 participants per group). 3 sessions (á 60 minutes) per week for 12 consecutive weeks
  Interventions: Behavioral: Physical exercise
- Cognitive-behavioral therapy (Active Comparator): Cognitive-behavioral therapy conducted in groups (5-8 participants per group). 1 session (á 2-2.25 hours depending on group size) per week for 12 consecutive weeks
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Physical exercise — Manualised Exercise performed in groups (5-8 participants per group). 3 sessions (á 60 minutes) per week for 12 consecutive weeks
  Arms: Physical exercise
Behavioral: Cognitive-behavioral therapy — Cognitive-behavioral therapy conducted in groups (5-8 participants per group). 1 session (á 2-2.25 hours depending on group size) per week for 12 consecutive weeks
  Arms: Cognitive-behavioral therapy

SUMMARY:
The purpose of this study is to compare manualised physical exercise conducted in groups to manualised cognitive-behavioral therapy conducted in groups as treatment for panic disorder with or without agoraphobia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Clinical diagnosis of panic disorder with and without agoraphobia according to The Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR, 4th ed., text revision; American Psychiatric Association, 2000), established through administration of Structural Clinical Interview for DSM-IV axis I disorders (SCID I; First, Spitzer, Gibbon, & Williams, 1995).

Exclusion Criteria:

* Brain-organic disorders according to DSM-IV-TR
* The presence of psychotic disorders according to DSM-IV-TR, established through administration of SCID I
* Present substance-abuse
* Medical condition that excludes participation in physical activity
* Major Depressive Disorder according to DSM-IV-TR established through administration of SCID I.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mobility Inventory (MI) - Alone & Accompanied | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up
Agoraphobic Cognitions Questionnaire (ACQ) | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up
Body Sensations Questionnaire | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up
Panic frequency - Self-report & Clinician-rating | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up
Panic distress/disability - Self-report & Clinician-rating | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up
State-Trait Anxiety Inventory - State & Trait (STAI S/T) | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up
Beck Depression Inventory II (BDI-II) | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up
Quality of Life Inventory (QoLI) | Baseline; Pre-treatment; Post-treatment; 6-months follow-up; 12-monthts follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anders Hovland, PsyD, Principal Investigator — University of Bergen
Locations (1):
- Solli Hospital, Bergen, Nesttun, Norway